CLINICAL TRIAL: NCT02695836
Title: Improving Nursing Home Care Through Feedback On PerfoRMance Data (INFORM)
Brief Title: Improving Nursing Home Care Through Feedback On PerfoRMance Data
Acronym: INFORM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Carole Estabrooks, Professor & Canada Research Chair in Knowledge Translation, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RES0026204; Application Number: 341532 (Other: Canadian Institute of Health Research - Open Operating Grant)
Record Dates: First submitted 2016-01-22; First posted 2016-03-01 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Organizational Context
Keywords: Audit and Feedback; Nursing Homes; Organizational Context; Quality Improvement; Care Aides; Leadership; Resident Assessment Instrument (RAI); Alberta Context Tool (ACT)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to study arm assignment
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard feedback (Active Comparator): Facilities in this arm will receive an initial face-to-face dissemination workshop that includes feedback of research data on modifiable aspects of their microsystem context but no goal setting.
  Interventions: Other: Initial face-to-face dissemination workshop
- Basic assisted feedback (Experimental): In addition to the face-to-face dissemination workshop, facilities in this arm will receive a face-to-face goal setting workshop focused on modifiable areas of their microsystem context and two virtual support workshops at six month intervals.
  Interventions: Other: Initial face-to-face dissemination workshop; Other: Face-to-face goal setting workshop; Other: Virtual support workshops
- Enhanced assisted feedback (Experimental): In addition to the face-to-face dissemination workshop, facilities in this arm will receive an additional face-to-face goal setting workshop focused on modifiable areas of their microsystem context, two additional face-to-face support workshops at six month intervals plus on-demand email and telephone support.
  Interventions: Other: Initial face-to-face dissemination workshop; Other: Face-to-face goal setting workshop; Other: Face-to-face support workshops; Other: On-demand email and telephone support

INTERVENTIONS:
Other: Initial face-to-face dissemination workshop — Managers and directors of care will receive a printed report (tailored to their facility) on their facility's performance and performance of each unit (microsystem) within that facility. The workshop will include a presentation of the feedback reports with a particular focus on the core set of actionable context targets (Formal Interactions, Evaluation, Social Capital, Organizational Slack (OS) - Time) in the face-to-face workshops. Following the presentation, participants will discuss their reports in facilitated, round-table group discussions to a) help with interpretation of the results overall, b) draw attention to elements of context that are modifiable, c) encourage microsystem teams to work on improving the more modifiable areas
Other: Face-to-face goal setting workshop — Sessions will build on the dissemination workshops and will be held three months after. Feedback reports on Formal Interactions, Evaluation, Social Capital, and Organizational Slack (OS) - Time will be discussed. Small group activities will take place including: a) reflecting on context data, b) performance goal setting using the 'tell and sell' method, which capitalizes on the workshop leaders' perceived expertise about what goals are achievable, c) establishing a series of proximal learning goals that will provide teams with explicit strategies for attaining performance goals set in (b). An action plan and instructions for reporting back at the Virtual Support Workshop will be provided.
  Arms: Basic assisted feedback; Enhanced assisted feedback
Other: Virtual support workshops — On virtual support workshop will be held six months after the feedback and goal setting workshop, and a second one another six months later. Groups will a) report on their progress in the proximal learning goals and strategies used toward their performance goals, b) discuss challenges they may be encountering, and c) receive support from the research team in addressing these challenges.
  Arms: Basic assisted feedback
Other: Face-to-face support workshops — On face-to-face support workshop will be held six months after the feedback and goal setting workshop, and a second one another six months later. Groups will a) report on their progress in the proximal learning goals and strategies used toward their performance goals, b) discuss challenges they may be encountering, and c) receive support from the research team in addressing these challenges. Workshops will be attended by all participating teams from a region, to maximize opportunities for teams to learn from one another and trouble-shoot together with the support of workshop leaders.
  Arms: Enhanced assisted feedback
Other: On-demand email and telephone support — Participants can contact the research team if needed with requests for support in defining or implementing improvement strategies or dealing with barriers towards improvement.
  Arms: Enhanced assisted feedback

SUMMARY:
This project will evaluate three different strategies to get research findings back to managers of care units in nursing homes. Feedback will be provided in a timely and effective way so that it results in improvements in organizational context (modifiable features of the care unit work environment, such as Formal Interactions, Informal Interactions, Social Capital or Slack Time), quality of care providers' work life (e.g., burnout, job satisfaction, general health) and quality of care. Three feedback packages will be tested to determine the strategy that is most effective at fostering improvements and is also cost-effective. The project will be carried out in nursing homes in Alberta and British Columbia. The information developed will contribute to better care for Canadian seniors who spend their final years in a nursing home.

DETAILED DESCRIPTION:
Background:

The purpose of this project is to systematically evaluate a tailored intervention targeting the leaders of clinical microsystems (care units) in residential long term care (nursing home - NH) settings. The intervention is designed to feedback performance data for improvement. This project is a key element of a long term program of research (Translating Research in Elder Care - TREC) focused on advancing knowledge translation science. TREC's goal is to improve quality of care, and in so doing, improve quality of life for older adults in NHs and work life for their care providers. TREC specifically focuses on the important role of organizational context (modifiable elements of the work environment) at the clinical microsystem (clinical unit) level in NHs.

Aims:

1. Evaluate and compare a standard feedback and 2 assisted, goal-directed feedback strategies
2. Assess sustainability and long term effects of each strategy
3. Refine a practical assisted feedback strategy for use in NHs targeting the leaders of clinical microsystems

Design: Pragmatic, three-arm, parallel, cluster-randomized trial; stratified permuted block randomization; baseline assessment, 1-year intervention period, post-intervention assessment and 1-year long-term follow up. NHs will be randomly assigned to Standard Feedback (SF), Basic Assisted Feedback (BAF) or Enhanced Assisted Feedback (EAF).

Setting: Stratified (region by size by operator) random sample of 67 eligible NHs from four regions in two provinces: Alberta (Edmonton, Calgary) and British Columbia (Fraser Health, Interior Health). Facilities participate in a longitudinal observational study (part of TREC) that generates a rich resident, staff, unit, and facility level database.

Random assignment: The cohort of 67 NHs is recruited. All sites have agreed to and expect standard feedback. 22 facilities (60 eligible units) were randomly assigned to SF, 22 facilities (70 eligible units) to BAF, and 23 facilities (73 eligible units) to EAF. Facilities assigned to BAF or EAF will be approached and offered additional feedback. Managers will be explained the specific extra feedback (treatment) they will receive, but they will be blinded to group allocation.

Sample: Target of the intervention are managers of the care units within the NHs. To avoid contamination effects, randomization will be done at the facility level, with all included unit managers of the same facility receiving the same feedback intervention. To determine sample size a computer simulation-based sample size approach was adapted that accounted for multiple repeated measures in three study arms, and the complex nested structure (time points nested within each care unit, and units clustered within facilities). Power and sample size were estimated based on a mixed-effects regression model. Using data from the previous phase of TREC (2007-2012) the required parameters to be entered into the model were estimated. Assumptions were that SF will increase the primary outcome (Formal Interactions [FI] score) by 0.2, BAF will increase the FI score by 0.4, and EAF will increase the FI score by 0.6. With an assumed power of 0.90, a significance level of 0.05 and an attrition rate of 25%, a total of 144 care units will be needed (48 NHs with an average number of three units or 72 NHs with an average number of two units).

Intervention:

All three groups will receive a face-to-face Dissemination Workshop (feedback of research data on modifiable aspects of the care unit context). The SF group will receive no additional intervention. The BAF and EAF arms will receive an additional face-to-face Goal Setting Workshop and two Support Workshops at six month intervals. Support Workshops will be virtual in the BAF arm and face-to-face in the EAF arm. In addition the EAF arm will receive on-demand email and phone support. Feedback will include data about four aspects of organizational context that are routinely measured in TREC with the validated Alberta Context Tool (ACT). Four of ten ACT concepts were selected for specific focus: 1) the number of Formal Interactions (FIs) care aides have with other providers and with patients/families; 2) the amount of Slack Time care aides have; 3) Evaluation (unit feedback) Practices, and 4) Social Capital. The intervention is designed to improve performance on these aspects of context. Intervention target is the clinical microsystem (clinical unit) managerial team within NHs: unit care managers and the director of care.

Primary outcome: Formal Interactions (FI), defined as formal exchanges through scheduled activities that can promote the transfer of knowledge (details see outcomes section). Previous research in TREC (2007-2012) clearly suggested that some context areas on the ACT have the potential to exert greater impact on quality of care and implementation of change. Of these, FI has the greatest single impact. At the microsystem level no unit scored above 1.9 (max. possible score is 4) and the mean was 1.3, leaving substantial room for improvement. The correlation of FI with the overall ACT context score is .5, and combinations of FI plus three additional ACT concepts (Evaluation, Social Capital, Slack Time) increased the correlation to .8. Field surveys suggested that care managers are interested in FI as an actionable concept of facility context and consider it a prime accessible target for action and change. FI constitutes the most actionable, cost-effective, and easy-to-improve context for enhancing quality, since the mechanisms for improvement are readily available. FI makes use of existing resources and requires little investment beyond organizational adaptations (scheduling training or meeting sessions, developing educational materials to disseminate research findings, etc.). Finally and importantly, FI is also a proximal goal. The organizational behavior literature is clear that the goal set cannot be too distal.

Secondary outcomes:

1. ACT context measures: Feedback, Social Capital, Organizational Slack - Time
2. Staff outcomes: research use, psychological empowerment, job satisfaction
3. Resident outcomes: quality indicators from the Resident Assessment Instrument - Minimum data Set 2.0 (RAI): worsening pain, declining behavioral symptoms. The RAI is used internationally for comprehensive geriatric assessment of the health, physical, mental, and functional status of NH. In Canada its use is mandated in several provinces/territories, as well as by the Canadian Institute of Health Information for national reporting.
4. Unit and facility outcomes: response to major near misses, managers' organizational citizenship behavior, performance reports, quality improvement activities

Process evaluations:

1. Workshop evaluation surveys
2. Intervention protocol checklists to evaluate fidelity of workshop delivery
3. Focus groups with managerial teams directly before the first support workshop and one month before the second support workshop
4. Cost accounting of the intervention

Statistical Analysis:

Primary Analysis: To compare the effectiveness of the three feedback interventions in improving the FI score, mixed-effects regression models will be used. The models will account for multiple measures within each unit and clustering of units within facilities. All analyses will be adjusted for the three stratification variables of the TREC facility sample (region, owner-operator model and facility size). Characteristics of units and facilities will be compared using descriptive statistics at baseline. Based on this, models will be adjusted for baseline variables that differ significantly between treatment groups. Data will be assessed whether they meet the assumptions of this model (multivariate normality, linearity, normally distributed, uncorrelated residuals, random effects with mean zero) and models will be adjusted accordingly. Intention-to-treat analysis will be conducted, as this best reflects the pragmatic nature of the study. These results will be compared to an as-treated analysis, which better reflects adherence/non-adherence with the intervention. Reporting of these findings will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

Secondary Analyses: Change of secondary outcomes (resident outcomes, i.e., RAI quality indicators, staff outcomes and organizational variables) will be monitored over time in each study arm, and outcomes will be compared between the three study arms using descriptive statistics, Statistical Process Control methods, and appropriate significance tests (t tests for normally distributed, linear, continuous outcomes; non-parametric tests for variables that don't meet these assumptions; chi tests for categorical outcomes). A dichotomous variable (improved/not improved) will be assigned to each unit in the intervention. Then, using logistic regression with improvement as the outcome the effects of context (using ACT scales), best practice use, and staff characteristics on improvement will be investigated. To this end a reliable classification system for individual control charts was developed.

ELIGIBILITY:
Facilities:

Inclusion Criteria:

* Participates in the Translating Research in Elder Care program
* Located in on of the following health regions in Alberta and British Columbia: Alberta North, Alberta South, Fraser Health, Interior Health
* At least one care unit in the facility with 10 or more care aide responses to our TREC survey
* Care aide responses can be assigned to a care unit in the facility as defined by TREC (TREC microsystem)

Exclusion Criteria:

* Does not participate in TREC
* Not located in the above named health regions
* No care unit in the facility with 10 or more care aide responses to our TREC survey
* Care aide responses cannot be assigned to a TREC defined microsystem

Care Units:

Inclusion Criteria:

* 10 or more care aide responses to our TREC survey
* Clearly identifiable unit leader (can also lead other units)
* Stable leadership over the last year

Exclusion Criteria:

* Less than 10 care aide responses to our TREC survey
* No clearly identifiable unit leader
* No stable leadership over the last year

Care Professionals:

Inclusion Criteria:

* Leader of one or more included care units (care managers, directors of care)
* Assistant leader of one or more included care units
* Quality improvement specialist or clinical educator/instructor of one or more included care units
* Employed in the facility
* Has been covering in this role on this unit for 1 year or more
* Leaders can bring care providers with no formal leadership or expert position (e.g., care aide, nurses, allied health providers) to the workshops

Exclusion Criteria:

* Not employed in the facility (e.g., casual)
* Has been covering in this role on this unit for less than 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Formal Interactions (FI) | Post-intervention assessment, up to 6 months (July-December 2017)
  FI is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "formal exchanges that occur between individuals working within an organization (unit) through scheduled activities that can promote the transfer of knowledge." FI includes four items asking care aides how often, in the last typical month, they participated in (a) team meetings about residents, (b) family conferences, (c) change-of-shift report, and (d) continuing education (conferences, courses) outside the nursing home (rated from 1=never to 5=almost always). To score FI, scores of each item are recoded (1 and 2 => 0; 3 => .5; 4 and 5 => 1) and summed up. FI therefore is scored with values ranging from 0 to 4, and averaged.
Formal Interactions (FI) | Long-term follow up, up to 6 months (January-June 2019)
  FI is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "formal exchanges that occur between individuals working within an organization (unit) through scheduled activities that can promote the transfer of knowledge." FI includes four items asking care aides how often, in the last typical month, they participated in (a) team meetings about residents, (b) family conferences, (c) change-of-shift report, and (d) continuing education (conferences, courses) outside the nursing home (rated from 1=never to 5=almost always). To score FI, scores of each item are recoded (1 and 2 => 0; 3 => .5; 4 and 5 => 1) and summed up. FI therefore is scored with values ranging from 0 to 4, and averaged.

SECONDARY OUTCOMES:
Evaluation (Unit Feedback) | Post-intervention assessment, up to 6 months (July-December 2017)
  Evaluation is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the process of using data to assess group/team performance and to achieve outcomes in organizations or units (i.e., evaluation)". Evaluation includes six items asking care aides to rate regular feedback activities on their care unit (e.g., if their team routinely monitors their performance with respect to previously generated action plans). The six items are rated on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Evaluation score, the six items are averaged.
Evaluation (Unit Feedback) | Long-term follow up, up to 6 months (January-June 2019)
  Evaluation is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the process of using data to assess group/team performance and to achieve outcomes in organizations or units (i.e., evaluation)". Evaluation includes six items asking care aides to rate regular feedback activities on their care unit (e.g., if their team routinely monitors their performance with respect to previously generated action plans). The six items are rated on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Evaluation score, the six items are averaged.
Social Capital | Post-intervention assessment, up to 6 months (July-December 2017)
  Social Capital is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the stock of active connections among people. These connections are of three types: bonding, bridging, and linking". Social Capital includes six items asking care aides to rate characteristics of their care team (e.g., if they are "comfortable talking about resident care issues with those in positions of authority"). The six items are rated on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Evaluation score, the six items are averaged.
Social Capital | Long-term follow up, up to 6 months (January-June 2019)
  Social Capital is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the stock of active connections among people. These connections are of three types: bonding, bridging, and linking". Social Capital includes six items asking care aides to rate characteristics of their care team (e.g., if they are "comfortable talking about resident care issues with those in positions of authority"). The six items are rated on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Evaluation score, the six items are averaged.
Organizational Slack (OS) Time | Post-intervention assessment, up to 6 months (July-December 2017)
  OS Time is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the cushion of actual or potential time resources which allows a care unit to adapt successfully to internal pressures for adjustments or to external pressures for changes". OS Time includes four items asking care aides to rate how often they have time to do certain things during resident care (e.g., "do something extra for residents"). The Items are rated on a 5-point Likert scale 1 = never to 5 = almost always. To obtain the OS Time score, the four items are averaged.
Organizational Slack (OS) Time | Long-term follow up, up to 6 months (January-June 2019)
  OS Time is one of ten concepts included in the Alberta Context Tool (ACT). It is defined as "the cushion of actual or potential time resources which allows a care unit to adapt successfully to internal pressures for adjustments or to external pressures for changes". OS Time includes four items asking care aides to rate how often they have time to do certain things during resident care (e.g., "do something extra for residents"). The Items are rated on a 5-point Likert scale 1 = never to 5 = almost always. To obtain the OS Time score, the four items are averaged.
Instrumental Research Use (IRU) | Post-intervention assessment, up to 6 months (July-December 2017)
  IRU is defined as "the use of observable research-based practices when caring for residents. Practice may be guided by guidelines, protocols, routines, care plans or procedures that are based on research". IRU includes one item asking care aides to rate how often on their last typical work day they used this type of research (best practices). The Item is rated on a 5-point Likert scale 1 = never to 5 = almost always.
Instrumental Research Use (IRU) | Long-term follow up, up to 6 months (January-June 2019)
  IRU is defined as "the use of observable research-based practices when caring for residents. Practice may be guided by guidelines, protocols, routines, care plans or procedures that are based on research". IRU includes one item asking care aides to rate how often on their last typical work day they used this type of research (best practices). The Item is rated on a 5-point Likert scale 1 = never to 5 = almost always.
Conceptual Research Use (CRU) | Post-intervention assessment, up to 6 months (July-December 2017)
  CRU is defined as "the cognitive, reflective use of research (best practices) where the best practice knowledge may change one's opinion or mind set about a specific practice area but not necessarily one's direct actions. It is an indirect application of research findings". CRU includes five items asking care aides to rate how often on their last typical work day research (best practice knowledge) did, for example, raise their awareness about new ways to care for residents. The Items are rated on a 5-point Likert scale 1 = never to 5 = almost always. To obtain the CRU score, the five items are averaged.
Conceptual Research Use (CRU) | Long-term follow up, up to 6 months (January-June 2019)
  CRU is defined as "the cognitive, reflective use of research (best practices) where the best practice knowledge may change one's opinion or mind set about a specific practice area but not necessarily one's direct actions. It is an indirect application of research findings". CRU includes five items asking care aides to rate how often on their last typical work day research (best practice knowledge) did, for example, raise their awareness about new ways to care for residents. The Items are rated on a 5-point Likert scale 1 = never to 5 = almost always. To obtain the CRU score, the five items are averaged.
Psychological Empowerment Scale | Post-intervention assessment, up to 6 months (July-December 2017)
  Psychological Empowerment reflects an active orientation in which an individual wishes and feels able to shape his or her work role and context. It is a state rather than a trait and is specific to the work domain (e.g. is not generalizable to one's life situations and roles). The Psychological Empowerment Scale includes twelve items that are scored on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. The twelve items reflect four different sub-scales - Meaning, Competence, Determination, and Impact - each of which is formed by three items. Each of the four sub-scale scores is obtained by averaging the respective three items.
Psychological Empowerment Scale | Long-term follow up, up to 6 months (January-June 2019)
  Psychological Empowerment reflects an active orientation in which an individual wishes and feels able to shape his or her work role and context. It is a state rather than a trait and is specific to the work domain (e.g. is not generalizable to one's life situations and roles). The Psychological Empowerment Scale includes twelve items that are scored on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. The twelve items reflect four different sub-scales - Meaning, Competence, Determination, and Impact - each of which is formed by three items. Each of the four sub-scale scores is obtained by averaging the respective three items.
Job Satisfaction (Michigan Organizational Assessment Questionnaire Job Satisfaction Subscale - MOAQ-JSS-3) | Post-intervention assessment, up to 6 months (July-December 2017)
  The MOAQ-JSS-3 is a global job satisfaction measure that reflects affective components (i.e. ones feelings about his/her job). It includes three items that are scored on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Job Satisfaction score, the three items are averaged.
Job Satisfaction (Michigan Organizational Assessment Questionnaire Job Satisfaction Subscale - MOAQ-JSS-3) | Long-term follow up, up to 6 months (January-June 2019)
  The MOAQ-JSS-3 is a global job satisfaction measure that reflects affective components (i.e. ones feelings about his/her job). It includes three items that are scored on a 5-point Likert scale from 1 = strongly disagree to 5 = strongly agree. To obtain the Job Satisfaction score, the three items are averaged.
Prevalence of Worsening Pain | Post-intervention assessment, up to 6 months (July-December 2017)
  This is one of 35 quality indicators that can be derived from the Resident Assessment Instrument - Minimum Data Set (RAI-MDS) 2.0, which is collected in quarterly assessments for all residents. Prevalence of Worsening Pain is one of 13 practice sensitive RAI-MDS 2.0 quality indicators (i.e., modifiable by care staff). It is based on the items J2a - Frequency of pain and J2b - Intensity of pain and reflects the percentage of residents with greater pain at target assessment relative to prior assessment.
Prevalence of Worsening Pain | Long-term follow up, up to 6 months (January-June 2019)
  This is one of 35 quality indicators that can be derived from the Resident Assessment Instrument - Minimum Data Set (RAI-MDS) 2.0, which is collected in quarterly assessments for all residents. Prevalence of Worsening Pain is one of 13 practice sensitive RAI-MDS 2.0 quality indicators (i.e., modifiable by care staff). It is based on the items J2a - Frequency of pain and J2b - Intensity of pain and reflects the percentage of residents with greater pain at target assessment relative to prior assessment.
Prevalence of Declining Behavioral Symptoms | Post-intervention assessment, up to 6 months (July-December 2017)
  This is one of 35 quality indicators that can be derived from the Resident Assessment Instrument - Minimum Data Set (RAI-MDS) 2.0, which is collected in quarterly assessments for all residents. Prevalence of Declining Behavioral Symptoms is one of 13 practice sensitive RAI-MDS 2.0 quality indicators (i.e., modifiable by care staff). It is based on the items E4a - Wandering, E4b - Verbally abusive, E4c - Physically abusive, E4d - Socially inappropriate behaviour, and reflects the percentage of residents who have declining behaviour symptoms. Where 1 or more of the indicators are greater at the target assessment than the prior assessment.
Prevalence of Declining Behavioral Symptoms | Long-term follow up, up to 6 months (January-June 2019)
  This is one of 35 quality indicators that can be derived from the Resident Assessment Instrument - Minimum Data Set (RAI-MDS) 2.0, which is collected in quarterly assessments for all residents. Prevalence of Declining Behavioral Symptoms is one of 13 practice sensitive RAI-MDS 2.0 quality indicators (i.e., modifiable by care staff). It is based on the items E4a - Wandering, E4b - Verbally abusive, E4c - Physically abusive, E4d - Socially inappropriate behaviour, and reflects the percentage of residents who have declining behaviour symptoms. Where 1 or more of the indicators are greater at the target assessment than the prior assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Carole A Estabrooks, PhD, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ginsburg LR, Hoben M, Easterbrook A, Anderson RA, Estabrooks CA, Norton PG. Fidelity is not easy! Challenges and guidelines for assessing fidelity in complex interventions. Trials. 2021 May 29;22(1):372. doi: 10.1186/s13063-021-05322-5. PMID 34051830
- [Derived] Hoben M, Ginsburg LR, Easterbrook A, Norton PG, Anderson RA, Andersen EA, Bostrom AM, Cranley LA, Lanham HJ, Weeks LE, Cummings GG, Holroyd-Leduc JM, Squires JE, Wagg AS, Estabrooks CA. Comparing effects of two higher intensity feedback interventions with simple feedback on improving staff communication in nursing homes-the INFORM cluster-randomized controlled trial. Implement Sci. 2020 Sep 10;15(1):75. doi: 10.1186/s13012-020-01038-3. PMID 32912323
- [Derived] Hoben M, Norton PG, Ginsburg LR, Anderson RA, Cummings GG, Lanham HJ, Squires JE, Taylor D, Wagg AS, Estabrooks CA. Improving Nursing Home Care through Feedback On PerfoRMance Data (INFORM): Protocol for a cluster-randomized trial. Trials. 2017 Jan 10;18(1):9. doi: 10.1186/s13063-016-1748-8. PMID 28069045
- See also: Translating Research in Elder Care (TREC) program — https://trecresearch.ca/
- See also: Improving Nursing Home Care through Feedback on PerfoRMance Data (INFORM) trial — https://trecresearch.ca/research/inform